CLINICAL TRIAL: NCT06212362
Title: Stepped Care Versus Group Cognitive Behaviour Therapy for Paediatric Anxiety in Primary Care: a Multisite Randomised Controlled Non-inferiority Trial
Brief Title: Stepped Care Versus Group Cognitive Behaviour Therapy for Paediatric Anxiety in Primary Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government); Vastra Gotaland Region (Other Government)
Responsible Party: Principal Investigator, Johan Åhlén, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: jaai02
Record Dates: First submitted 2023-12-26; First posted 2024-01-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Anxiety
Keywords: anxiety; children; cognitive behavioural therapy
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Multi-site randomised non-inferiority trial. Half of the participants will be randomised to receive Step-by-step, and half of participants will be randomised to receive Cool Kids.
Who Masked: Outcomes Assessor
Masking Description: Assessors conducting 12 weeks-assessments will be blind to treatment allocation. The outcome measure (PARS) is identical for both groups, ensuring that the assessors remain blind. At the 12 week-assessment, participants will be reminded to not reveal their arm allocation. To measure blinding integrity, all assessors will record whether the participating families inadvertently reveal their group allocation, and subsequently guess each participant's treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Step-by-Step treatment (Experimental)
  Interventions: Behavioral: Step-by-step
- Cool Kids treatment (Active Comparator)
  Interventions: Behavioral: Cool Kids

INTERVENTIONS:
Behavioral: Step-by-step — The Step-by-Step follows a stepped care approach, were all children (and caregivers) complete the first step (a brief group intervention followed by an individual session). Those with more needs are offered to continue to step 2 where individual CBT is given.
  Step 1 Session 1-4: Group sessions including psychoeducation, parenting skills and mapping stress and vulnerability factors, exposure and coping skills (90 minutes) Session 5: Individual session - If ending after step 1 a maintenance plan is completed. If continuing to step 2 continued exposure and selection of optional focus areas such as emotion regulation, social skills, stress- and vulnerability factors, child worry or parental worry. (45 minutes)
  Step 2 Session 6-8: Individual sessions - Exposure and selected focus areas. (45 minutes)
  Arms: Step-by-Step treatment
Behavioral: Cool Kids — The Cool Kids Program is an Australian manualized group CBT treatment of child anxiety, which has been broadly implemented in Sweden. Several studies have found evidence of its efficacy.
  Session 1-10: Group sessions including psychoeducation, cognitive restructuring (gather evidence to reevaluate anxiety related thoughts), parent skills, exposure, social skills, coping skills (cognitive and behavioral strategies to handle anxiety reactions, learning problem-solving skills). (90-120 minutes)
  Arms: Cool Kids treatment

SUMMARY:
Objectives: Over the past decade in Sweden, a novel approach to primary healthcare units, known as first-line mental health (FLMH), has been introduced to enhance mental health services for children and adolescents. Through a structured and collaborative method involving experts, clinicians, and patients, a trans-diagnostic psychological intervention for anxiety was formulated based on cognitive behavioural therapy (CBT), designed to align with the FLMH care framework. This study seeks to assess the efficacy of the CBT intervention "Step-by-Step" in a randomised, single-blind, parallel-group, multisite non-inferiority trial. The objective is to investigate whether this treatment is not less effective than the evidence-based Cool Kids program.

Rationale for the Study: Childhood anxiety is prevalent and linked to suffering and impairment across various life domains. While cognitive behavioural therapy (CBT) is a proven treatment for anxiety disorders in children, there is a pressing need to enhance access to such interventions. Introducing CBT for childhood anxiety within primary care settings offers an avenue for early and readily available treatment. However, a gap exists in the availability of CBT interventions specifically designed for and assessed within primary care contexts.

DETAILED DESCRIPTION:
BACKGROUND: Anxiety is the primary reason for contacting the First Line Mental Health (FLMH) in Sweden. Urgently needed is the increased accessibility of evidence-based interventions (EBIs) for child and adolescent anxiety. Cognitive behavioural therapy (CBT) has proven efficacy in child anxiety treatment, though predominantly within psychiatric settings. The FLMH focuses on early interventions for mild to moderate mental health problems in children and adolescents, posing a challenge in identifying EBIs adapted to their needs. The FLMH services often struggle with fitting full-length EBIs into primary care or, more commonly, shorten interventions without empirical support for maintained efficacy. A structured co-creative approach was used to develop a CBT intervention, "Step-by-step," for FLMH. Preliminary testing indicated acceptability, appropriateness, and feasibility, with positive feedback leading to minor revisions in the treatment manual.

OBJECTIVE: The overarching aim of this research project is to increase the availability of evidence-based psychological treatments for children with anxiety treated within primary care.

PRIMARY RESEARCH QUESTION: Is Step-by-step an effective and resource efficient treatment in reducing anxiety severity compared to an evidence-based and well-established treatment (Cool Kids).

SECONDARY RESEARCH QUESTIONS: Is Step-by-step more suitable for certain subgroups of patients in terms of baseline characteristics? Is Step-by-step non-inferior to the Cool Kids regarding children's depressive symptoms, and quality of life? Is Step-by-step non-inferior to the Cool Kids in reducing family accommodation and increasing parental self-efficacy? Are changes in family accommodation and parental self-efficacy mediators of treatment effects? Are there differences in mental health care utilisation between treatments (three-year follow up of health care registers)? Do Step-by-step and Cool Kids differ in terms of treatment adherence, patient satisfaction, and therapists' fidelity? Do Step-by-step and Cool Kids fit the needs of patients?

PROJECT DESCRIPTION: Half of the participants will be randomised to receive Step-by-step, and half of participants will be randomised to receive Cool Kids. All participants will be followed up 12 weeks after treatment initiation (post assessment), and one year after the post assessment. The primary endpoint is set to the post assessment. Participants will be asked to consent for linkage with registers, including retrieving information about utilization of health care up to three years after the post assessment.

CONTROL GROUP JUSTIFICATION: The researchers opted for Cool Kids as the comparator in order to assess and compare the effectiveness of the new treatment, Step-by-Step, against an established evidence-based treatment. Further, the Cool Kids is the most implemented treatment for childhood anxiety in Sweden. Finally, waitlist would not be an ethical choice because there are efficient treatment options available for anxiety in children.

POWER ANALYSIS: The researchers found one previous paediatric anxiety treatment trial employing a non-inferiority design with the Pediatric Anxiety Rating Scale (PARS) as the primary outcome. In this trial, researchers used six points as non-inferiority margin. However, given that the standard deviation of the PARS typically varies between 5-6 and treatment effects for clinician rated outcome (CBT vs. controls) on average are equivalent to a Cohen's d of 0.94, a 6 points margin is likely too large.

Preliminary results from a study exploring the minimal clinical individual difference (MCID) on PARS benchmarked against the Clinical Global Impression Scale (CGI) suggested a change of 6 points as MCID between pre- and post-treatment. We used simulated data with a pre- post within subject design to explore different non-inferiority margins' effect on the proportions of individuals meeting the MCID criteria. Compared to a change on the PARS corresponding to approximately 70% meeting the MCID criteria (i.e., parallel to remission rates in previous trials of the Cool Kids), a change of 3 points less, would correspond to approximately 50% meeting the MCID criteria.

Given the information above, we decided to set the non-inferiority margin to 3 points. The non-inferiority analysis will be based on the PARS scores at the primary endpoint (12 weeks after treatment initiation).

We estimated the statistical power for different sample sizes that the Step-by-step is not worse than the Cool Kids at the 12-week post assessment. We considered one time-point and a response rate of 90%. The estimated power was the observed rejection proportion over 10,000 generated simulated datasets. The data were generated based on the information available in a pilot study on 30 patients. Based on the simulation, the estimated enrolment of participants is set to 154 participants. In other words, if the Step-by-step is truly non-inferior to the Cool Kids program, 154 patients will give an estimated probability of more than 90% that the upper limit of a one-sided 97.5% confidence interval will be below the non-inferiority limit of 3 points on the PARS. No specific non-inferiority margin is defined for the secondary outcome measures.

SCREENING AND RECRUITMENT: At first visit (face-to face, by video or telephone) at the FLMH-unit, the therapist typically collects information about the medical history (including potential previous mental health problems) of the child, assess the severity of mental distress and the global function of the child. On this occasion, eligible children and parents/guardians will receive oral and written information about the study and will be given an opportunity to ask questions about participation. If interested in participation, informed consent will be obtained from all parents/guardians (digitally). If not interested in participation, patients will be offered regular care at the FLMH-unit. In cases where the child needs contact with specialised psychiatric care and/or other organisations than FLMH (i.e., social services or school) families will be referred according to standard routines at the FLMH units.

Children with parents/guardians' consent will be interviewed with the PARS by a FLMH-therapist. During the PARS interview, children and parents/guardians will complete additional baseline assessment via the secure online data collection tool. After the PARS interview, the therapist will assess adherence to the inclusion criteria, and carefully evaluate potential exclusion criteria to ensure that participants meet the required eligibility standards for enrolment in the study. Upon confirming a participant's eligibility for inclusion in the study, the therapist will proceed to open a sequentially numbered envelope. These envelopes have been meticulously prepared in advance by a researcher and contain the randomised assignment.

RANDOMISATION, ENROLMENT AND MASKING: Participants will be randomised at a 1:1 ratio to Step-by-step or Cool Kids. Randomisation and masking procedures will be conducted by an external researcher not involved in the recruitment. For each semester, all FLMH-units will receive 14 sealed envelopes (numbered between 1-14) with seven Step-by-step and seven Cool Kids allocations. We will use a block-randomisation, with block sizes randomly varying of 2 and 4. The randomisation will be generated using a computer random number generator by the researchers. Assessors conducting post- and follow-up assessments will be blind to treatment allocation. The outcome measure (PARS) is identical for both groups, ensuring that the assessors remain blind. At post- and follow-up assessments, participants will be reminded not to reveal their arm allocation. To measure blinding integrity, all assessors will record whether the participating families inadvertently reveal their group allocation, and subsequently guess each participant's treatment allocation.

END OF TRIAL: The trial will end when the registry data (at the 3-year follow up) has been collected.

STATISTICAL ANALYSES: Data will be analysed according to intention-to-treat principles and according to per protocol as adequate in non-inferiority trials. Data analysis on the continuous outcome measures will be performed with mixed-effect regression analyses for repeated measures. The model will include fixed effects of time, treatment group, and an interaction effect of treatment group by time, as well as random intercept to account for individual differences. Ordinal data will be analysed with ordinal regression, binary data will be analysed with logistic regression. Within- and between-group effect sizes will be reported as Cohen's d.

DATA MANAGEMENT All aspects of data management of the trial will comply with the General Data Protection Regulation and good clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* The child is 7-12 years old (Confirmed by the parent/guardian and from medical records)
* The child suffers from mild to moderate anxiety. The term "mild to moderate anxiety" has not been explicitly defined but is a term aimed to specify a demarcation between the FLMH and the psychiatric specialist services. Adequate level of care for the patient is decided based on an overall clinical assessment. The Children Global Assessment Scale (CGAS) is often used to guide the decision on level of care, where a CGAS value above 60 clearly indicates primary care services, a value below 50 clearly indicates specialist services. For values between 50 and 60 the overall clinical evaluation of symptom severity and impaired function guide the decision on level of care. (Confirmed by the assessor at the FLMH-unit).

Exclusion Criteria:

* Other psychiatric or developmental disorders than anxiety, or social issues that primarily require other interventions, i.e., where an intervention targeting mild to moderate anxiety is not adequate. (Confirmed by assessor at the FLMH-unit).
* The child has another ongoing psychological intervention. An ongoing psychological treatment for any other psychiatric disorder. (Confirmed by the parent/guardian).

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in Pediatric Anxiety Rating Scale, PARS (clinician rated) | Three timepoints: Baseline assessment, 12 weeks after treatment initiation (post assessment), and 12 months after the post assessment
  The PARS is a semi-structured clinical interview aimed to assess the severity and functional impairment of anxiety in children aged 6-17 years. Questions are asked to both children and parents. The ratings of severity and impairment is made based on the overall picture of anxiety symptoms. PARS has been used as an outcome measure in several treatment studies.

SECONDARY OUTCOMES:
Change in Child Anxiety Severity Scale, CASS) (child- and parent-rated) | Four timepoints: Baseline assessment, 5 weeks after treatment initiation (mid-treatment assessment), 12 weeks after treatment initiation (post assessment), and 12 months after the post assessment
  The CASS is a six-item self-rated (or parent-rated) questionnaire, and is an adapted version of the clinician-rated PARS that aims to assess the severity of anxiety associated with common anxiety disorders. It is rated on a 3-point Likert scale (or 5-point Likert scale for parents) with higher scores indicating more anxiety. The self-rated version has been adapted and translated by our research group, and we have an ongoing study where we will evaluate the psychometric properties in a clinical sample and a school sample.
Change in The Revised Children's Anxiety and Depression Scale, RCADS (child- and parent-rated) | Three timepoints: Baseline assessment, 12 weeks after treatment initiation (post assessment), and 12 months after the post assessment
  The RCADS is a validated scale that aims to assess the frequency of anxious and depressive symptoms. Items are rated on a 4-point Likert scale with higher scores indicating more anxiety or depression. Parents and children will complete the brief 25-item RCADS.
Change in The Family Accommodation Scale - Anxiety, FASA-A (child- and parent-rated) | Four timepoints: Baseline assessment, 5 weeks after treatment initiation (mid-treatment assessment), 12 weeks after treatment initiation (post assessment), and 12 months after the post assessment
  The FASA-A is a validated self-rated (or parent-rated) questionnaire of the parent's accommodation to the child's anxiety, including 13 items (each item scored on a Likert scale between 0-4 where higher scores indicate more accommodation)
Change in the Child Health Utility 9D, CHU9D (parent-rated) | Three timepoints: Baseline assessment, 12 weeks after treatment initiation (post assessment), and 12 months after the post assessment
  CHU9D is a parent-rated questionnaire of the child's quality of life, including 9 items, each scored 1-5 where lower scores indicate better quality of life.
Change in Brief Parental Self-Efficacy, BPSES (parent-rated) | Four timepoints: Baseline assessment, 5 weeks after treatment initiation (mid-treatment assessment), 12 weeks after treatment initiation (post assessment), and 12 months after the post assessment
  BPSES is a brief questionnaire consisting of five questions designed to measure parental self-efficacy. Items are rated on a 5-point Likert scale, where higher scores indicate self-efficacy. BPSES was originally developed to be useful in the context of parenting support for parents of children with conduct problems. In this study, researchers use a version of BPSES customised towards parenting support for children with anxiety.

OTHER OUTCOMES:
Unintended Treatment Effects | 12 weeks after treatment initiation (post assessment)
  Parents will be asked to answer four questions on whether they experienced any unintended treatment effects, the nature of the effect(s), how they affected the child and/or the parent during treatment and after treatment
Mental Health Care (register data) | Three years following the completion of treatment
  The number of care visits, psychiatric diagnoses, and psychotropic medication use in inpatient and outpatient child and adolescent psychiatric care, as well as care for mental health issues in primary care, will be collected from administrative healthcare registers.
Treatment Adherence (clinician-rated) | 12 weeks after treatment initiation (post assessment)
  Therapists will report attendance to sessions (yes/no) and additionally rate engagement in treatment based on parents/guardians' verbal reports on their compliance with homework assignments and other behaviors consistent with the treatment plan. Therapists will make one overall rating for the whole treatment ranging from 1 (Not at all engaged in home assignment or an equally relevant activity) to 5 (Highly engaged, exceeding expectations, in home assignment or an equally relevant activity)
The Client Satisfaction Questionnaire, CSQ-8 (parent-rated) | 12 weeks after treatment initiation (post assessment)
  The CSQ is a self-rated scale with 8 items measuring different aspects of satisfaction with treatment, e.g., perception of quality of treatment, if the treatment adequately addressed their needs and overall satisfaction
Treatment fit to participants need (interview with parents) | 12 weeks after treatment initiation (post assessment)
  The interview guide focuses on parents' treatment experience, expectations, assessment of treatment suitability for their child's needs, the decision-making process to discontinue or proceed to step 2, collaboration with the therapist, and potential feedback for improving the treatment model. The interview is estimated to take approximately 45 to 60 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Åhlén, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Solna, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Some information collected in the research project (survey data and clinician assessments) may be shared with national and international collaborators within the EU/EEA and in the USA. The transfer will apply to studies with similar research questions as in the current project, such as meta-analyses that combine results from multiple studies. The transferred personal data will be coded and done in accordance with the applicable legislation at any given time. Relevant agreements will be established in cases required by current legislation. Recipients in third countries must handle personal data with the same level of protection as within the EU.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Available on request after the results are published in peer-reviewed journal.
Access Criteria: Each request will be assessed individually